CLINICAL TRIAL: NCT05078125
Title: ECG and CMR for Predicting PVCs in Cardiomyopathic Patients
Brief Title: Electrocardiographic and Cardiac Magnetic Resonance Predictors of Ventricular Arrhythmias in Cardiomyopathic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Mohamed Aly, Resident doctor of cardiology .Luxor International Hospital, Assiut University
Other Study IDs: AssiutU KMAly
Record Dates: First submitted 2021-10-02; First posted 2021-10-14 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Premature Ventricular Complex
MeSH Terms: conditions — Ventricular Premature Complexes | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Holter monitoring — 24 hours Holter monitoring

SUMMARY:
This study aims to assess ECG changes for predicting ventricular arrhythmia in cardiomyopathic patients

DETAILED DESCRIPTION:
This study aims to assess ECG markers based on 24-hour Holter ECG recordings for predicting ventricular arrhythmia in patients with Structural Heart disease who have left ventricular dysfunction and Left Ventricular Ejection Fraction ≤40%. With special concerns to underlying structural abnormalities in cardiomyopathic patients using Cardiac Magnetic Resonance to determine ventricular function, scar distribution, and grey zone analysis

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic and non-ischemic cardiomyopathy, EF < 40 %
* Patient haemodynamically stable
* Patients accept to make test

Exclusion Criteria:

1. Patients with underlying arrhythmia ex heart block or atrial arrhythmia like PACs, AF.
2. Patients on arrhythmogenic drugs ex digitalis, amiodarone.
3. Patients on underlying Pacemaker device or CRT-D.
4. Patients with MI in less than 40 days
5. Patients refuse to make test .

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study is anticipated to include all consecutive eligible cardiomyopathic patients.
Sampling Method: Probability Sample
Enrollment: 79 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Twenty-four hours Holter monitoring after Magnetic Resonance Imaging | One year
  24 Holter monitoring to detect PVCs burden which is defined as ≥10% of total beats

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mathew T, Williams L, Navaratnam G, Rana B, Wheeler R, Collins K, Harkness A, Jones R, Knight D, O'Gallagher K, Oxborough D, Ring L, Sandoval J, Stout M, Sharma V, Steeds RP; British Society of Echocardiography Education Committee. Diagnosis and assessment of dilated cardiomyopathy: a guideline protocol from the British Society of Echocardiography. Echo Res Pract. 2017 Jun;4(2):G1-G13. doi: 10.1530/ERP-16-0037. PMID 28592613
- [Result] Pinto YM, Elliott PM, Arbustini E, Adler Y, Anastasakis A, Bohm M, Duboc D, Gimeno J, de Groote P, Imazio M, Heymans S, Klingel K, Komajda M, Limongelli G, Linhart A, Mogensen J, Moon J, Pieper PG, Seferovic PM, Schueler S, Zamorano JL, Caforio AL, Charron P. Proposal for a revised definition of dilated cardiomyopathy, hypokinetic non-dilated cardiomyopathy, and its implications for clinical practice: a position statement of the ESC working group on myocardial and pericardial diseases. Eur Heart J. 2016 Jun 14;37(23):1850-8. doi: 10.1093/eurheartj/ehv727. Epub 2016 Jan 19. PMID 26792875
- [Result] Sharma E, Arunachalam K, Di M, Chu A, Maan A. PVCs, PVC-Induced Cardiomyopathy, and the Role of Catheter Ablation. Crit Pathw Cardiol. 2017 Jun;16(2):76-80. doi: 10.1097/HPC.0000000000000106. PMID 28509708
- [Result] Lee DC, Markl M, Dall'Armellina E, Han Y, Kozerke S, Kuehne T, Nielles-Vallespin S, Messroghli D, Patel A, Schaeffter T, Simonetti O, Valente AM, Weinsaft JW, Wright G, Zimmerman S, Schulz-Menger J. The growth and evolution of cardiovascular magnetic resonance: a 20-year history of the Society for Cardiovascular Magnetic Resonance (SCMR) annual scientific sessions. J Cardiovasc Magn Reson. 2018 Jan 31;20(1):8. doi: 10.1186/s12968-018-0429-z. PMID 29386064